CLINICAL TRIAL: NCT04644315
Title: A Phase II, Open-Label, Single Arm Decentralized Home-Based Approach Study to Evaluate the Efficacy and Safety of Alectinib in Locally-Advanced or Metastatic ALK-Positive Solid Tumors
Brief Title: A Home-Based Approach Study to Evaluate the Efficacy and Safety of Alectinib in Locally-Advanced or Metastatic ALK-Positive Solid Tumors
Acronym: ALpha-T
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The data from this study is no longer needed.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO41929
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms; Colorectal Neoplasms; Melanoma; Pancreatic Neoplasms; Sarcoma; Ovarian Neoplasms; Brain Neoplasms; Thyroid Neoplasms; Neuroendocrine Tumors; Cholangiocarcinoma; Salivary Gland Neoplasms; Head and Neck Neoplasms; Thyroid Cancer, Papillary; Lymphoma, Large-Cell, Anaplastic; Neoplasms by Site; Respiratory Tract Neoplasms; Thoracic Neoplasms; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Central Nervous System
Keywords: agnostic; ALK+; Alk-positive; ALK positive; ALK mutation; GI; breast; sarcoma; neuroendocrine; female reproductive; ALK; ALK fusions; ALK gene rearrangements; colorectal cancer; entrectinib; basket study; salivary gland cancers; primary brain tumors; melanoma; sarcomas; papillary thyroid cancer; renal cell cancer; pancreatic cancer; breast cancer; cholangiocarcinoma; head & neck cancers; ovarian cancer; anaplastic lymphoma kinase positive; solid tumors; ALK+ solid tumors
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Melanoma; Pancreatic Neoplasms; Sarcoma; Ovarian Neoplasms; Brain Neoplasms; Thyroid Neoplasms; Neuroendocrine Tumors; Cholangiocarcinoma; Salivary Gland Neoplasms; Head and Neck Neoplasms; Thyroid Cancer, Papillary; Lymphoma, Large-Cell, Anaplastic; Neoplasms by Site; Respiratory Tract Neoplasms; Thoracic Neoplasms; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Carcinoma, Renal Cell; Breast Neoplasms | interventions — alectinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALK-positive Solid Tumors (Experimental): Participants with locally advanced or metastatic ALK-positive tumors will receive alectinib twice daily (BID) until disease progression, unacceptable toxicity, death, or withdrawal from the study for any reason.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive 600 mg oral alectinib BID until disease progression, unacceptable toxicity, withdrawal from treatment, or death.
  Other Names: Alecensa

SUMMARY:
This study will evaluate the efficacy and safety of alectinib in participants with Anaplastic Lymphoma Kinase (ALK)-positive locally advanced or metastatic solid tumors other than lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ALK-positive locally-advanced or metastatic solid tumor excluding lung cancer
* ALK-positive tumor as per Foundation Medicine, Inc (FMI) next-generation sequencing (NGS) (NGS F1CDx, F1LCDx, or F1HEME) or per local accredited laboratory using validated NGS testing of tumor tissue or peripheral blood
* No alternative effective standard therapy available, or standard therapy considered unsuitable or intolerable to the participant
* Other cancer therapies are allowed, including investigational drugs, if any treatment-related toxicities (excluding alopecia) have resolved to grade </= 1 or to laboratory values as defined by the protocol
* Measurable disease at baseline as assessed by the Investigator per RECIST v1.1 or RANO criteria (for participants with primary CNS tumors)
* Life expectancy of at least 12 weeks
* Eastern cooperative oncology group (ECOG) performance status of 0-2
* Adequate hemataologic, hepatic, and renal function
* Participants with primary central nervous system (CNS) tumors are available
* Participants with brain or leptomeningeal metastasis are allowed in the study if asymptomatic and if they meet additional criteria as defined by the protocol
* Willingness to comply with study procedures
* Willingness to comply with home-base approach and visits by Mobile Nurses
* Ability to swallow alectinib capsules intact
* Women of childbearing potential must test negative for pregnancy at screening and prior to the first dose of study drug
* Women of childbearing potential must agree to remain abstinent or use contraceptive methods as defined by the protocol and refrain from donating eggs during the treatment period and for at least 90 days after the last dose of alectinib
* Men must agree to remain abstinent or use contraceptive methods as defined by the protocol and refrain from donating sperm during the treatment period and for at least 90 days after the last dose of alectinib

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of alectinib
* Lung Cancer
* Patients with one of the following ALK point mutations: I1171X, G1202R, V1180L
* Prior therapy with an ALK inhibitor
* Liver disease as described in the protocol
* Known HIV, hepatitis B, or hepatitis C (HCV) infection
* Patients with symptomatic bradycardia
* Patients with symptomatic or unstable brain metastasis; patients with primary CNS tumors are allowed
* Malabsorption syndrome or any other condition that would interfere with enteral absorption
* Incomplete recovery from any surgery prior to treatment
* Any other malignancies within 5 years prior to enrollment, except for those described in the protocol
* Any serious medical condition or abnormality in clinical laboratory tests that, in the Investigator's judgment, precludes the patient's safe participation in and completion of the study
* History of hypersensitivity to any of the ingredients in the alectinib drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (29):
  - Science 37, Inc, Culver City, California
  - Science 37-Basem; Dept 004- Basem, Culver City, California
  - Science 37-Beg; Dept 001 Dr. M. Beg, Culver City, California
  - Science 37-Cannon; Dept 002-Cannon, Culver City, California
  - Science 37-Kurzrock; Dept 005-Kurzrock, Culver City, California
  - Science 37-Thomas; Dept 006-Thomas, Culver City, California
  - Homebased Telemedicine, Los Angeles, California
  - Homebased Telemedicine, Sacramento, California
  - Homebased Telemedicine, San Diego, California
  - Homebased Telemedicine, San Francisco, California
  - Homebased Telemedicine, San Jose, California
  - Homebased Telemedicine, Jacksonville, Florida
  - Homebased Telemedicine, Miami, Florida
  - Homebased Telemedicine, Orlando, Florida
  - Homebased Telemedicine, Tampa, Florida
  - Homebased Telemedicine, Fort Wayne, Indiana
  - Homebased Telemedicine, Indianapolis, Indiana
  - Homebased Telemedicine, Minneapolis, Minnesota
  - Homebased Telemedicine, Saint Paul, Minnesota
  - Homebased Telemedicine, St Louis, Missouri
  - Homebased Telemedicine, Buffalo, New York
  - Homebased Telemedicine, New York, New York
  - Homebased Telemedicine, Philadelphia, Pennsylvania
  - Homebased Telemedicine, Pittsburgh, Pennsylvania
  - Homebased Telemedicine, Austin, Texas
  - Homebased Telemedicine, Dallas, Texas
  - Homebased Telemedicine, Houston, Texas
  - Homebased Telemedicine, Richmond, Virginia
  - Homebased Telemedicine, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- ALK-positive Solid Tumors: Participants with locally advanced or metastatic ALK-positive tumors were to receive alectinib twice daily (BID) until disease progression, unacceptable toxicity, death, or withdrawal from the study for any reason.
Period: Overall Study
Arm/Group | ALK-positive Solid Tumors
Started | 1
Completed | 0
Not Completed | 1
Not completed — Subject withdrawal of consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The risk of participant re-identification is unacceptable for a population of n=1 and this value will therefore not be provided.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The risk of participant re-identification is unacceptable for a population of n=1 and this value will therefore not be provided.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The risk of participant re-identification is unacceptable for a population of n=1 and this value will therefore not be provided.

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) as Determined by the Investigator Per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Time Frame: Approximately 1 year
Population: Confirmed ORR was defined as the proportion of participants with a complete or partial response (CR or PR) confirmed at least 28 days after initial response.
Measure: Number; unit: Percentage
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 1
Percentage | 0

2. Secondary Outcome: Confirmed ORR as Determined by Blinded Independent Center Review (BICR) Per RECIST v1.1
Time Frame: 0 days
Population: BICR was not performed.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR) as Determined by Both the Investigator and by BICR Per RECIST v1.1
Time Frame: From first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 5 years)
Population: DOR was defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause and could not be calculated due to an insufficient number of participants with the event.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival (PFS) as Determined by Both the Investigator and by BICR Per RECIST v1.1
Time Frame: From first dose of alectinib to disease progression or death from any cause, whichever occurs first (up to 5 years)
Population: PFS was defined as the time from the first dose of alectinib to disease progression or death from any cause and could not be calculated due to an insufficient number of participants with the event.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

5. Secondary Outcome: Central Nervous System (CNS) ORR by BICR Per RECIST v1.1
Time Frame: Baseline up to 5 years
Population: CNS ORR was defined as the objective tumor response rate (CR or PR) of CNS lesions and could not be calculated due to an insufficient number of participants with the event.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

6. Secondary Outcome: CNS DOR by BICR Per RECIST v1.1
Time Frame: From the first observation of CNS response to the first observation of CNS progression or death from any cause (up to 5 years)
Population: CNS DOR was defined as the time from the first observation of CNS response until the first observation of CNS progression or death from any cause and could not be calculated due to an insufficient number of participants with the event.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival (OS)
Time Frame: From the first dose of study drug to death from any cause (up to 5 years)
Population: OS was defined as the time from first dose of study drug to death from any cause- and could not be calculated due to an insufficient number of participants with the event.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Approximately 1 year
Measure: Number; unit: Percentage
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 1
Percentage | 100

9. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Time Frame: Approximately 1 year
Measure: Number; unit: Percentage
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 1
Percentage | 100

10. Secondary Outcome: Plasma Concentration of Alectinib
Time Frame: Baseline up to 5 years
Population: Plasma concentration data was not collected as the data for one participant was not sufficient.
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

11. Secondary Outcome: ORR in Participants With Primary CNS Tumors as Determined by Both BICR and the Investigator Per Response Assessment in Neuro-Oncology (RANO) Criteria
Time Frame: Up to 5 years
Population: as for outcome 5
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

12. Secondary Outcome: DOR in Participants With Primary CNS Tumors as Determined by Both BICR and the Investigator Per RANO Criteria
Time Frame: as for outcome 3
Population: as for outcome 3
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

13. Secondary Outcome: PFS in Participants With Primary CNS Tumors as Determined by Both BICR and the Investigator Per RANO Criteria
Time Frame: From first dose of alectinib to disease progression or death from any cause, whichever occurs first (up to 5 years)
Population: as for outcome 4
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

14. Secondary Outcome: OS in Participants With Primary CNS Tumors
Time Frame: From the first dose of study drug to death from any cause (up to 5 years)
Population: as for outcome 7
Arm/Group | ALK-positive Solid Tumors
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Arm/Group | ALK-positive Solid Tumors
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK-positive Solid Tumors (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK-positive Solid Tumors (N=1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight decreased (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04644315/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04644315/SAP_001.pdf